CLINICAL TRIAL: NCT03812731
Title: Incidence of Urethrocutaneous Fistula Following Distal Hypospadias Repair With and Without Caudal Epidural Block - A Pilot Study
Brief Title: Incidence of Urethrocutaneous Fistula With and Without Caudal Epidural Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, Dr Nitin Sethi, Associate Professor & Consultant, Sir Ganga Ram Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EC/01/19/1478
Record Dates: First submitted 2019-01-19; First posted 2019-01-23 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Distal Hypospadias
MeSH Terms: interventions — Ropivacaine; Fentanyl

STUDY DESIGN:
Intervention Model Description: 30 male patients aged 1-8 years, ASA physical status I/II, and undergoing distal hypospadias repair will be randomly allocated to one of the following two groups:
  GROUP I- (Caudal group, n= 15) Children will receive general anesthesia (GA) and analgesia will be maintained with caudal epidural block (CEB) with 0.2% ropivacaine:1 ml/kg.
  GROUP II- (Non-caudal group, n= 15) Children will receive general anaesthesia (GA) and analgesia will be maintained with intravenous fentanyl citrate 1mcg/kg/hr.
  roup-1 [CLADS Group, n=60]: Anaesthesia will be induced and maintained with propofol administered using the BIS feedback-based automated CLADS. Group-2 [Desflurane Group, n=60]: Anaesthesia will be induced with propofol CLADS and will be maintained intraoperatively by Desflurane titrated to BIS monitoring.
Who Masked: Participant, Outcomes Assessor
Masking Description: The attending anaesthesiologist will not be blinded to the technique utilised to administer GA. An independent assessor blinded to the technique of GA will follow up the patients to determine the incidence of uretherocutaneous fistula
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caudal Group (Active Comparator): Children will receive oral midazolam 0.25 mg/kg thirty minutes before induction. Inhalational induction will be carried with incremental concentration of sevoflurane upto 8% in 50% oxygen and nitrous oxide mixture. As soon as the child will be asleep, ASA standard monitors (SPO2, HR, ECG and NIBP) will be attached. Intravenous access with age appropriate IV cannula will be secured. Injection fentanyl citrate 2 mcg/ kg followed by injection atracurium 0.5 mg/kg will be administered. Appropriate size LMA Pro SealTM will be inserted and pressure controlled ventilation will be instituted.
  Children in will then receive CEB with 0.2 % ropivacaine 1-ml/kg for maintaining analgesia
  Interventions: Drug: Ropivacaine
- Non- Caudal Group (Active Comparator): Children will receive oral midazolam 0.25 mg/kg thirty minutes before induction. Inhalational induction will be carried with incremental concentration of sevoflurane upto 8% in 50% oxygen and nitrous oxide mixture. As soon as the child will be asleep, ASA standard monitors (SPO2, HR, ECG and NIBP) will be attached. Intravenous access with age appropriate IV cannula will be secured. Injection fentanyl citrate 2-mcg/ kg followed by injection atracurium 0.5 mg/kg will be administered. Appropriate size LMA Pro SealTM will be inserted and pressure controlled ventilation will be instituted.
  Children in will then receive fentanyl citrate 1-mcg/kg/hr for maintaining analgesia
  Interventions: Drug: Fentanyl Citrate

INTERVENTIONS:
Drug: Ropivacaine — Intraoperatively after induction of anaesthesia caudal epidural block will be administered with 0.2% ropivacaine 1-ml/kg
  Arms: Caudal Group
Drug: Fentanyl Citrate — Intraoperatively after induction of anaesthesia fentanyl 1-mcg/kg/hour will be administered
  Arms: Non- Caudal Group

SUMMARY:
The study is designed to explore any association between the caudal epidural block(CEB) given for perioperative analgesia and the occurrence of urethrocutaneous fistula postoperatively in children undergoing distal hypospadias repair .We also intend to study the duration of penile engorgement due to CEB causing penile oedema which may subsequently play a role in fistula formation. The pilot study will recruit children under 8 years of age diagnosed with distal hypospadias scheduled to undergo Tubularised Incised Plate Urethroplasty, operated by a single paediatric surgeon. General anaesthesia will be induced with sevoflurane in oxygen nitrous oxide mixture supplemented by fentanyl citrate and atracurium besylate in all children. LMA Pro SealTMof appropriate size will be inserted. Children in group I will then be given caudal epidural block (CEB) as per our practice protocol. Children in group II will be given additional intravenous fentanyl citrate. All children will be followed postoperatively till 3 months to evaluate incidence of urethtocutaneous fistula. The prospective study attempts to eliminate previously reported confounding factors.

DETAILED DESCRIPTION:
CEB is routinely used along with general anaesthesia for inguinal and genital surgeries. It provides intraoperative and postoperative analgesia, is safe, simple and has success rate of more than 90% in children.It decreases the requirement of inhalational anaesthetics and narcotics, decreases stress hormone release and facilitates early recovery. Hypospadias is the most common congenital anomaly of penis, incidence being 1 in 300 live births. Hypospadias repair is a technical procedure that can be associated with significant complications such as meatal stenosis, stricture, glans dehiscence and flap necrosis Urethrocutaneous fisula formation is the most common complication after primary repair with an incidence of upto 20%. There have been controversies regarding the association of CEB with urethrocutaneous fistula. Some studies have reported a high incidence of postoperative urethrocutaneous fistula in children who received CEB while others have not confirmed any such relationship. Association between urethrocutaneous fistula and site of urethral opening, age of patient, duration of surgery, surgeon's expertise, use of subcutaneous epinephrine and use of preoperative testosterone has been found. Penile engorgement, post inflammatory response and tissue oedema may be contributory factors for development of fistula. However any association between CEB and fistula formation is not clear. All studies, except one, are retrospective, limited by small sample size and presence of various confounding factors. The present study is aimed to explore any association between CEB and urethrocutaneous fistula. The study will be conducted in children with distal hypospadias only; they will be operated by a single surgeon, without the use of subcutaneous epinephrine, so that any association, if at all between CEB and urethrocutaneous fistula becomes evident.

ELIGIBILITY:
Inclusion Criteria:

1. Male children l
2. 1 to 8 years of age
3. ASA physical status I and II
4. Distal hypospadias -

Exclusion Criteria:

1. Simultaneously undergoing any other procedure
2. Local infection in sacral region
3. Bleeding diathesis
4. Preoperative testosterone stimulation

Ages: 1 Year to 8 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Only male patients with distal hypospadias will be included
Enrollment: 30 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2019-11-28 (Actual)

PRIMARY OUTCOMES:
Incidence of urethrocutaneous fistula | From one day after surgery(0-hours, baseline) till 3-months post surgery
  Patients undergoing distal hypospadias repair will be followed up for occurrence of uretherocutaneous fistula

SECONDARY OUTCOMES:
Penile Engorgement | After induction of anaesthesia (0-hours, baseline) till end of surgery
  Length of penis from pubic bone to glans tip and mid shaft circumference i.e. girth around the widest part of the penile shaft will be calculated
Changes in intra-operative heart rate (beats per minute) | From beginning of anesthesia (0-hours, baseline) till 2-hours intraoperatively
  Comparison of intra-operative heart rate between both the arms will be done
Change in Intra-operative blood pressure - systolic , diastolic, and mean (mmHg) | rom beginning of anesthesia (0-hours, baseline) till 2-hours intraoperatively
  Comparison of intra-operative blood pressure- systolic, diastolic, and mean between both the arms will be done
Postoperative analgesia requirement | From end of anaesthesia (0-hours, baseline) till 24-hours postoperatively
  Additional fentanyl citrate 0.5-mcg/kg will be administered intravenously if the Face, Legs, Activity, Cry, Consolability scale (FLACC scale) score is > 3 and total amount administered will be recorded
Incidence of complications | From end of anaesthesia (0-hours, baseline) till 3-months postoperatively
  Complications of surgery such as infection, bleeding , hematoma, glans dehiscence, skin or flap necrosis will be noted

CONTACTS AND LOCATIONS:
Overall Officials: Deepali Shukla, DA, Principal Investigator — Sir Ganga Ram Hospital; Archna Koul, MS, MCH, Study Director — Sir Ganga Ram Hospital
Locations (1):
- Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No